CLINICAL TRIAL: NCT01092780
Title: An Active-Comparator Controlled Single Dose Study to Evaluate the Pharmacodynamics/Efficacy of MK-7288 in Sleep Apnea Patients
Brief Title: Pharmacodynamics and Efficacy of MK-7288 in Adults With Sleep Apnea (MK-7288-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7288-010; MK-7288-010 (Other: Merck study number)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Apnea, Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — MK-7288; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil (Experimental): Participants received single doses of study drug in the following order: MK-7288 10 mg in Treatment Period 1, Placebo (Pbo) in Treatment Period 2, MK-7288 20 mg in Treatment Period 3 and Modafinil 200 mg in Treatment Period 4. The first 3 treatment periods were followed by a 7-day washout period.
  Interventions: Drug: MK-7288; Drug: Placebo to MK-7288; Drug: Modafinil; Drug: Placebo to modafinil
- MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo (Experimental): Participants received single doses of study drug in the following order: MK-7288 20 mg in Treatment Period 1, MK-7288 10 mg in Treatment Period 2, Modafinil 200 mg in Treatment Period 3 and Placebo in Treatment Period 4. The first 3 treatment periods were followed by a 7-day washout period.
  Interventions: Drug: MK-7288; Drug: Placebo to MK-7288; Drug: Modafinil; Drug: Placebo to modafinil
- Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg (Experimental): Participants received single doses of study drug in the following order: Modafinil 200 mg in Treatment Period 1, MK-7288 20 mg in Treatment Period 2, Placebo in Treatment Period 3 and MK-7288 10 mg in Treatment Period 4. The first 3 treatment periods were followed by a 7-day washout period.
  Interventions: Drug: MK-7288; Drug: Placebo to MK-7288; Drug: Modafinil; Drug: Placebo to modafinil
- Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg (Experimental): Participants received single doses of study drug in the following order: Placebo in Treatment Period 1, Modafinil 200 mg in Treatment Period 2, MK-7288 10 mg in Treatment Period 3 and MK-7288 20 mg in Treatment Period 4. The first 3 treatment periods were followed by a 7-day washout period.
  Interventions: Drug: MK-7288; Drug: Placebo to MK-7288; Drug: Modafinil; Drug: Placebo to modafinil

INTERVENTIONS:
Drug: MK-7288 — one or two 10 mg capsules, orally, single dose
Drug: Placebo to MK-7288 — one or two capsules, orally, single dose
Drug: Modafinil — two 100 mg tablets, orally, single dose
  Other Names: PROVIGIL®
Drug: Placebo to modafinil — two 100 mg tablets, orally, single dose

SUMMARY:
This is a study of the safety and efficacy of MK-7288 for the treatment of excessive daytime sleepiness (EDS) in participants with obstructive sleep apnea (OSA)/hypopnea syndrome (HS) who are compliant with effective nasal continuous positive airway pressure (nCPAP) therapy. The goal of this study is to determine the effect of MK-7288 after single dose administration on promoting wakefulness as measured by sleep latency on Maintenance of Wakefulness Tests, and on driving performance as measured by standard deviation of lane position in simulated driving (country vigilance driving).

ELIGIBILITY:
Inclusion Criteria:

* Female participants are of non-child-bearing potential.
* Male participants who have female partner(s) of child-bearing potential must agree to use a medically acceptable method of contraception during the study.
* Participant has an International Classification of Sleep Disorders diagnosis of Obstructive Sleep Apnea/Hypopnea Syndrome.
* Participant has excessive daytime sleepiness.
* Participant has been using nCPAP treatment for at least 2 months.
* Participant reported total sleep time of >6 hours on at least 4 out of 7 nights each week
* Participant is willing to stay at the sleep laboratory for 5 overnight stays.
* Participant is willing to limit caffeine and alcohol consumption during the study.
* Participant has a valid driver's license in the past 5 years and has had at least 1 year of driving experience within the past 3 years.
* Participant's regular bedtime is between 9:00 p.m. and 12:00 a.m.

Exclusion Criteria:

* Participant has a history of cancer.
* Participant has any history of a significant neurological disorder.
* Participant has moderate or severe persistent asthma.
* Participant has a history of any of the following sleep disorders: narcolepsy, primary insomnia, Circadian rhythm sleep disorder, shift work sleep disorder, parasomnia including nightmare disorder, sleep terror disorder, rapid eye movement (REM) behavioral disorder, and sleepwalking disorder, periodic limb movement disorder, or restless leg syndrome.
* Participant consumes more than 10 cigarettes a day or routinely smokes during the night.
* Participant, in the opinion of the investigator, has a history or current evidence of any condition, therapy, lab abnormality or circumstances that might confound the results of the study, or interfere with participation for the full duration of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sun H, MacLeod C, Mostoller K, Mahon C, Han L, Renger JJ, Ma J, Brown KR, Schulz V, Kay GG, Herring WJ, Lines C, Rosen LB, Murphy MG, Wagner JA. Early-stage comparative effectiveness: randomized controlled trial with histamine inverse agonist MK-7288 in excessive daytime sleepiness patients. J Clin Pharmacol. 2013 Dec;53(12):1294-302. doi: 10.1002/jcph.182. Epub 2013 Oct 4. PMID 24122944

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 14 | 15 | 14 | 13
Completed | 14 | 15 | 14 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 14 | 15 | 14 | 13
Completed | 13 | 14 | 14 | 13
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Noncompliance with nCPAP | 1 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 13 | 14 | 14 | 13
Completed | 13 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 13 | 14 | 14 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Period: Treatment Period 3
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | MK-7288 10mg/Pbo/MK-7288 20mg/Modafinil | MK-7288 20mg/MK-7288 10mg/Modafinil/Pbo | Modafinil/MK-7288 20mg/Pbo/MK-7288 10mg | Pbo/Modafinil/MK-7288 10 mg/MK-7288 20mg
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All participants who were randomized in the study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (7.7) [32 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Sleep Latency Score on the Maintenance of Wakefulness Test (MWT) for Participants Taking MK-7288 Versus Placebo
Description: Study drug was administered at 08:00. MWT, an objective measure of the participant's ability to maintain wakefulness, was administered at 09:00, 11:00, 13:00 and 15:00. A least squares (LS) mean of the 4 MWTs performed at 09:00, 11:00, 13:00 and 15:00 was calculated. Latency for each MWT is defined as the time to onset of the first 16 continuous seconds of any stage of sleep; if no sleep has been observed according to these rules, then the latency is defined as 30 minutes. A higher MWT value is considered a better outcome.
Time Frame: 1, 3, 5 and 7 hours post dose
Population: The Per-Protocol (PP) population consisted of all participants who were compliant with the protocol and had available data from at least one treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Groups:
- MK-7288 10 mg: Participants received single doses of MK-7288 10 mg.
- MK-7288 20 mg: Participants received single doses of MK-7288 20 mg.
- Modafinil 200 mg: Participants received single doses of Modafinil 200 mg.
- Placebo: Participants received single doses of Placebo.
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Minutes | 18.66 [16.54 to 20.79] | 18.62 [16.50 to 20.73] | 20.71 [18.57 to 22.85] | 10.50 [8.35 to 12.65]
Statistical Analysis 1: Comparison: MK-7288 10 mg vs Placebo; Difference in least squares (LS) means; Test type: Superiority or Other; Difference in LS means = 8.16, 95% CI 2-sided [6.11 to 10.20]
Statistical Analysis 2: Comparison: MK-7288 20 mg vs Placebo; Difference in LS means; Test type: Superiority or Other; Difference in LS means = 8.11, 95% CI 2-sided [6.07 to 10.15]

2. Primary Outcome: Mean Score on Standard Deviation of Lane Position (SDLP) Driving Test for Participants Taking MK-7288 Versus Placebo
Description: Study drug was administered at 08:00. Driving performance was measured by the SDLP test which is a 45-minute driving simulation country vigilance test and was performed by participants at 10:00, 12:00 and 14:00. An LS mean of the 2 SDLP driving test results performed at 10:00 and 14:00 was calculated. A lower value is considered a better outcome.
Time Frame: 2, 4 and 6 hours post dose
Population: The PP population consisted of all participants who were compliant with the protocol and had available data from at least one treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Meters | 0.31 [0.28 to 0.35] | 0.32 [0.28 to 0.35] | 0.32 [0.29 to 0.36] | 0.39 [0.36 to 0.42]
Statistical Analysis 1: Comparison: MK-7288 10 mg vs Placebo; Difference in LS means; Test type: Superiority or Other; Difference in LS means = -0.07, 95% CI 2-sided [-0.10 to -0.05]
Statistical Analysis 2: Comparison: MK-7288 20 mg vs Placebo; Difference in LS means; Test type: Superiority or Other; Difference in LS means = -0.07, 95% CI 2-sided [-0.09 to -0.05]

3. Primary Outcome: Number of Participants Experiencing Clinical and Laboratory Adverse Events (AEs)
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the study drug, is also an AE.
Time Frame: Up to 36 days
Population: All Participants as Treated (APaT) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Participants
  Clinical AE | 30 | 37 | 16 | 12
  Laboratory AE | 1 | 1 | 0 | 1

4. Secondary Outcome: Mean Sleep Latency Score on the MWT for Participants Taking MK-7288 Versus Modafinil
Description: as for outcome 1
Time Frame: 1, 3, 5 and 7 hours post dose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Minutes | 18.66 [16.54 to 20.79] | 18.62 [16.50 to 20.73] | 20.71 [18.57 to 22.85] | 10.50 [8.35 to 12.65]
Statistical Analysis 1: Comparison: MK-7288 10 mg vs Modafinil 200 mg; Difference in LS means; Test type: Superiority or Other; Difference in LS means = -2.05, 90% CI 2-sided [-3.76 to -0.35]
Statistical Analysis 2: Comparison: MK-7288 20 mg vs Modafinil 200 mg; Difference in LS means; Test type: Superiority or Other; Difference in LS means = -2.10, 90% CI 2-sided [-3.79 to -0.40]

5. Secondary Outcome: Mean Sleep Latency Score on the MWT for Participants Taking Modafinil Versus Placebo
Description: as for outcome 1
Time Frame: 1, 3, 5 and 7 hours post dose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Minutes | 18.66 [16.54 to 20.79] | 18.62 [16.50 to 20.73] | 20.71 [18.57 to 22.85] | 10.50 [8.35 to 12.65]
Statistical Analysis 1: Comparison: Modafinil 200 mg vs Placebo; Test type: Superiority or Other; Difference in LS means = 10.21, 90% CI 2-sided [8.49 to 11.92]

6. Secondary Outcome: Mean Score on SDLP Driving Test for Participants Taking Modafinil Versus Placebo
Description: as for outcome 2
Time Frame: 2, 4 and 6 hours post dose
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Meters
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Number analyzed (Participants) | 54 | 55 | 53 | 52
Meters | 0.31 [0.28 to 0.35] | 0.32 [0.28 to 0.35] | 0.32 [0.29 to 0.36] | 0.39 [0.36 to 0.42]
Statistical Analysis 1: Comparison: Modafinil 200 mg vs Placebo; Difference in LS means; Test type: Superiority or Other; Difference in LS means = -0.07, 90% CI 2-sided [-0.08 to -0.05]

ADVERSE EVENTS:
Time Frame: Up to 36 days (Up to 3-4 days after last dose of study drug)
Description: The APaT population consisted of all participants who received at least one dose of study drug.
Arm/Group | MK-7288 10 mg | MK-7288 20 mg | Modafinil 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/55 | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 24/54 | 29/55 | 12/53 | 5/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7288 10 mg (N=54) | MK-7288 20 mg (N=55) | Modafinil 200 mg (N=53) | Placebo (N=52)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7288 10 mg (N=54) | MK-7288 20 mg (N=55) | Modafinil 200 mg (N=53) | Placebo (N=52)
Eructation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 6 (7) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 16 (16) | 16 (18) | 5 (5) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 10 (10) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.